CLINICAL TRIAL: NCT05071690
Title: COVID-19: Why Are Children Less Affected
Brief Title: Observational Study of Infants Fed on DHA (Breast Source or Milk Formula Source ) and Its Effects on Covid-19 Infected Infants and Severity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Collaborators: Faculty of medicine kafr elshiekh university (Unknown)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Clinical Scientist, Ministry of Health, Saudi Arabia
Other Study IDs: Observational COVID-19 Study
Record Dates: First submitted 2021-10-01; First posted 2021-10-08 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: DHA as Antioxidant Anti-inflammatory Immunomodulation , Overcome Cytokine Storm
Keywords: breast milk, Algae, DHA, cytokine storm, infant
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: on breast milk 50 baby full-term and infant follow up for covid-19 symptoms and measurement of plasma DHA
- arm 2: 50 baby depend on DHA source like infant formula milk or supplement with DHA

SUMMARY:
Observational Study of Infants Fed on DHA (Breast Source or Milk Formula Source ) and Its Effect on COVID-19 Severity

* Amr kamel khalil Ahmed ( drmedahmed@gmail.com ) Director of tuberculosis program Ghubera, public health department ,First health cluster ,Ministry of health , Riyadh, Saudia Arabia https://orcid.org/0000-0003-3477-236X
* Mahmoud Elkazzaz ( mahmoudramadan2051@yahoo.com ) Department of chemistry and biochemistry, Faculty of Science, Damietta University, Egypt https://orcid.org/0000-0003-3703-520X

Abstract

The novel SARS-CoV-2, which causes the disease called COVID-19, has rapidly spread across the globe. A striking and consistent observation has been the difference in severity of COVID-19 at different ages: severity, the need for hospitalization and mortality rise steeply with older age while severe disease and death are relatively rare in children and young adults. Most infants and children infected with SARS-CoV-2 are asymptomatic or have mild symptoms, most commonly fever, cough, pharyngitis, gastrointestinal symptoms and changes in sense of smell or taste. Whether infants and children are also less often infected by SARS-CoV-2 is an ongoing debate. Large epidemiological studies suggest that infants and children comprise only 1 to 2% of all SARS-CoV-2 cases. However, these numbers heavily depend on testing criteria and, in many reports, testing was done only in individuals who were symptomatic or required hospitalization, which is less often the case for children. Some studies suggest that infants and children are just as likely as adults to become infected with SARS-CoV-2.9 However, more recent studies report that children are less likely to get infected after contact with a SARS-CoV-2-positive individual.10-14 It has been suggested that children and adolescents have similar viral loads and may therefore be as likely to transmit SARS-CoV-2 as adults. In addition, the viral load may be similar in asymptomatic and symptomatic individuals. However, reassuringly, transmission in schools from children either to other children or to adults has been rare. The observation that children are less often infected with SARS-CoV-2 and that they have less severe symptoms is similar to that reported for SARS-CoV-1 and Middle East respiratory syndrome (MERS)-CoV. However, this pattern is strikingly different to that for infection with most other respiratory viruses (eg, respiratory syncytial virus (RSV), metapneumovirus, parainfluenza or influenza viruses), for which the prevalence and severity are both higher in children.Dr Amr kamel khalil Ahmed and Dr. Mahmoud Elkazzaz, the lead investigators of this observational study , recently published a preprint that demonstrated Docosahexaenoic acid (DHA) had a high binding affinity and greatest interactions with ACE2 active sites, as well as a moderate binding affinity and moderate interactions with the active sites of IL-6. The Docosahexaenoic acid (DHA) interacts with different active sites of IL6 and ACE2 which are involved in direct or indirect contacts with the ACE2 and IL-6 receptors which might act as potential blockers of functional ACE2 and IL-6 receptor complex. Docosahexaenoic acid (DHA) was detected in abundance in breast milk and other algal sources milk supplement used for newborns and children's feeding. As a result, we believe that docosahexaenoic acid (DHA) may protect children and newborns thorough competing with COVID-19 for ACE2 receptors and inhibiting IL-6 activity and may possibly help them avoid a cytokine storm and save their lives through inhibiting IL-6 and preventing SARS-CoV-2 RBD attachment to ACE2

DETAILED DESCRIPTION:
the study observational study case control study two groups of infants and children on DHA supplement A arm group on breast milk and measure the DHA level and determine the degree of severity of covid-19 symptoms according the classification of CDC the B arm infants on DHA at milk formula or DHA supplement and measure the DHA level and determine the severity of covid-19 according the classification of CDC

ELIGIBILITY:
Inclusion Criteria:

* full term baby infants and children until 5 years breast feeding or milk formula or supplement on DHA

Exclusion Criteria:

* above 5 years no congenital diseases outside kingdom saudia arabia preterm

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all preterm baby and infants and children under 5 years on breat mil or milk formula or DHA supplement
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
the severity of COVID-19 symptoms at infants and children on DHA at milk formula and on breast feeding | 6 month
  comparison between two control groups infants and children on breast milk and group on milk formula nouriched at DHA
measurement of percentage of plasma DHA at two groups of infants and children's | 6 month
  plasma DHA is very important to be measured

SECONDARY OUTCOMES:
THE duration of symptoms at two groups | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Amr K Ahmed, Principal Investigator — Ministry of Health, Saudia Arabia; Mahmoud R Elkazzaz, M.Sc of Biochemistry, Principal Investigator — Faculty of science Damietta university
Locations (2):
- Mahmoud, Kafr ash Shaykh, Kafr Elshiekh, Egypt
- Ministry of health.First health cluster ,Riaydh, Riyadh, Saudi Arabia